CLINICAL TRIAL: NCT00879216
Title: A Single Centre, Double-blind, Placebo Controlled Crossover Study in Elderly Male Subjects to Investigate the Plarmacodynamic Interaction of VA106483 Administered Concomitanctly With Alpha-blocker Therapy
Brief Title: VA106483 and Alpha Blocker Interaction Study in Elderly Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vantia Ltd (Industry)
Responsible Party: Medical Director, Charles River Clinical Services, Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 483-003
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Nocturia
Keywords: Nocturia; Hyptotension; Elderly; Males
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo
- VA106483 (Experimental)
  Interventions: Drug: VA106483

INTERVENTIONS:
Drug: VA106483 — 4 mg orally on either Day 7 or 10 with the placebo crossover treatment on the alternate day.
  Arms: VA106483
Drug: Placebo — 4 mg orally on either Day 7 or 10 with the placebo crossover treatment on the alternate day.
  Arms: Sugar pill

SUMMARY:
The main purpose of this study is to investigate whether the hypotensive effects of an alpha-blocker are increased when VA106483 is given at the same time.

DETAILED DESCRIPTION:
VA106483 is intended to be used as a treatment for patients suffering from nocturia (defined as waking to urinate at least once per night between periods of sleep). Nocturia is a condition that often worsens as sufferers get older. This may be due to an over-active bladder muscle, the bladder being able to hold less urine at night-time or over production of urine in the bladder at night. Some of the treatments available for nocturia have side-effects which make them unsuitable for elderly patients. These side-effects have not been seen in studies with VA106483, which makes it potentially suitable for treating elderly patients.

Nocturia is commonly associated with Benign Prostatic Hypertrophy (or BPH, a non-cancerous enlargement of the prostate gland, which often results in problems passing water). Of the patients who suffer from BPH, an estimated 40-85% experience the symptoms of waking at night to pass water.

Treatments which are commonly prescribed for BPH include alpha-blockers which work by improving urine flow by a muscle relaxant effect. Alpha-blockers are known to cause hypotension (lowering of blood pressure which can cause dizziness in some patients) . Since it is likely that subjects may be co-prescribed VA106483 and alpha-blockers, the purpose of this study is to determine that giving VA106483 does not increase the hypotensive effects of alpha-blockers

ELIGIBILITY:
Inclusion Criteria:

* Male aged 65 years of age and above
* No clinically important abnormal physical, laboratory or vital sign findings in the opinion of the Investigator
* Provision of written informed consent to participate
* No recent alpha-blocker therapy
* Not taking any concomitant medication known to be a cytochrome 3A4 inhibitor
* Not taking any prescribed or over the counter medications unless agreed with the Investigator and Sponsor
* No evidence of serious pathology or disease including poorly controlled endocrine disorders; active liver or biliary disease or severe kidney problems; syndrome of inappropriate antidiuretic hormone secretion
* No history of orthostatic hypotension or syncope.
* No known hypersensitivity to the IMP or alpha blocker, including severe lactose intolerance.
* No history of drug or alcohol abuse
* Negative for HIV, hepatitis B or C

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Blood pressure, Heart rate | For 8 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Charles River Clinical Services, Edinburgh, UK
Locations (1):
- Charles River Clinical Services, Edinburgh, United Kingdom